CLINICAL TRIAL: NCT00037778
Title: Genetic Modifiers of Cystic Fibrosis: Sibling Study
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1178; R01HL068927 (NIH)
Record Dates: First submitted 2002-05-20; First posted 2002-05-21 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Lung Diseases; Cystic Fibrosis
MeSH Terms: conditions — Lung Diseases; Cystic Fibrosis

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to identify modifier genes in cystic fibrosis (CF).

DETAILED DESCRIPTION:
BACKGROUND:

CF is a highly variable but inevitably fatal single gene disorder. Several lines of evidence suggest that genetic background contributes to the variability of cystic fibrosis phenotypes. The study will develop CF as a model for the identification of modifier genes by capitalizing on the availability of a large motivated population of affected twins and siblings.

The study is in response to a Request for Applications titled "Genetic Modifiers of Single Gene Defect Diseases" released in August 2000 and co-sponsored by the National Institute of Diabetes, Digestive, and Kidney Diseases.

DESIGN NARRATIVE:

The study has four aims: 1. To identify heritable CF phenotypes by twin study. Intrapair and interpair variance will be determined for selected CF phenotypes, and interclass correlations (monozygotic versus dizygotic) will be performed to identify CF phenotypes with a substantial heritable component. 2. To determine the contribution of genetic and other factors to the variability of CF phenotypes by analysis of affected sibs. Variance component methods will be used to evaluate the CF phenotypes that appear to be heritable based upon other studies or the results of aim 1. 3. To identify biologic phenotypes that correlate with heritable CF phenotypes by clinical study of twins and sibs. Multivariate analysis will be used to find biologic phenotypes associated with CF phenotypes. 4. To identify modifier genes and loci responsible for heritable CF phenotypes by linkage approaches. Identity by descent and transmission disequilibrium methods will be used to test linkage between candidate genes/loci and heritable CF phenotypes. To identify novel loci, genome-wide scans will be performed upon sib pairs selected for extreme concordance or discordance for heritable traits.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CF

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Siblings with cystic fibrosis
Sampling Method: Probability Sample
Enrollment: 3459 (Actual)
Dates: Start 2001-09; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Variation among genes in siblings with cystic fibrosis as assessed by DNA | Single collection

CONTACTS AND LOCATIONS:
Overall Officials: Garry Cutting, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

REFERENCES:
- [Background] McWilliams R, Hoover-Fong J, Hamosh A, Beck S, Beaty T, Cutting G. Problematic variation in local institutional review of a multicenter genetic epidemiology study. JAMA. 2003 Jul 16;290(3):360-6. doi: 10.1001/jama.290.3.360. PMID 12865377
- [Background] Groman JD, Hefferon TW, Casals T, Bassas L, Estivill X, Des Georges M, Guittard C, Koudova M, Fallin MD, Nemeth K, Fekete G, Kadasi L, Friedman K, Schwarz M, Bombieri C, Pignatti PF, Kanavakis E, Tzetis M, Schwartz M, Novelli G, D'Apice MR, Sobczynska-Tomaszewska A, Bal J, Stuhrmann M, Macek M Jr, Claustres M, Cutting GR. Variation in a repeat sequence determines whether a common variant of the cystic fibrosis transmembrane conductance regulator gene is pathogenic or benign. Am J Hum Genet. 2004 Jan;74(1):176-9. doi: 10.1086/381001. Epub 2003 Dec 18. PMID 14685937
- [Background] Boyle MP. Nonclassic cystic fibrosis and CFTR-related diseases. Curr Opin Pulm Med. 2003 Nov;9(6):498-503. doi: 10.1097/00063198-200311000-00009. PMID 14534402
- [Background] Hefferon TW, Groman JD, Yurk CE, Cutting GR. A variable dinucleotide repeat in the CFTR gene contributes to phenotype diversity by forming RNA secondary structures that alter splicing. Proc Natl Acad Sci U S A. 2004 Mar 9;101(10):3504-9. doi: 10.1073/pnas.0400182101. Epub 2004 Mar 1. PMID 14993601